CLINICAL TRIAL: NCT01981291
Title: Duration of Subgluteal Sciatic Nerve Block After Intra- or Perineural Injection of Mepivacaine: a Randomized, Controlled Trial
Brief Title: Duration of Sciatic Nerve Block After Injection of Local Anesthetic In or Around the Nerve
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Marco Baciarello, Assistant Professor, Anesthesia, Critical Care and Pain Medicine, University of Parma
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANEST-ORT-03
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Orthopedic Surgical Procedures; Postoperative Pain
Keywords: Lower Extremity; Sciatic Nerve; Anesthesia, Regional; Anesthetics, Local; Mepivacaine; Ultrasonography
MeSH Terms: conditions — Pain, Postoperative | interventions — Passive Cutaneous Anaphylaxis; Mepivacaine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perineural (Active Comparator): Patients in this group will receive a perineural injection of mepivacaine for subgluteal sciatic nerve block, in addition to a femoral nerve block and patient-controlled postoperative analgesia.
  Interventions: Procedure: Perineural Injection for Subgluteal Sciatic Nerve Block; Procedure: Femoral Nerve Block; Procedure: Patient-controlled postoperative analgesia; Drug: Mepivacaine
- Intraneural (Experimental): Patients in this group will receive an intraneural injection of mepivacaine for subgluteal sciatic nerve block, in addition to a femoral nerve block and patient-controlled postoperative analgesia.
  Interventions: Procedure: Intraneural Injection for Subgluteal Sciatic Nerve Block; Procedure: Femoral Nerve Block; Procedure: Patient-controlled postoperative analgesia; Drug: Mepivacaine

INTERVENTIONS:
Procedure: Intraneural Injection for Subgluteal Sciatic Nerve Block — The injection will start as the needle penetrates the outermost discernible layer of the nerve (epineurium) under ultrasound guidance. The injection will be adjudicated as "intraneural" if nerve cross section expansion and a reduction in echogenicity are observed.
  Short-axis real-time ultrasound imaging will be used, with an in-plane needle approach.
  Other Names: Injection beneath the common investing external layer; Subepineural Injection; Gluteal sciatic nerve block; Subparaneural injection
  Arms: Intraneural
Procedure: Perineural Injection for Subgluteal Sciatic Nerve Block — The injection will start as the needle indents the outermost discernible layer of the nerve (epineurium) under ultrasound guidance. The injection will be adjudicated as "intraneural" if the drug infiltrates the space between the epimysium of the surrounding muscles and the outer epineurium of the sciatic nerve.
  Short-axis real-time ultrasound imaging will be used, with an in-plane needle approach.
  Other Names: Injection outside the common investing external layer; Epineural injection; Extraneural injection
  Arms: Perineural
Procedure: Femoral Nerve Block — Patients will receive an ultrasound-guided femoral nerve block using a short- or long-acting local anesthetic, as deemed indicated.
Procedure: Patient-controlled postoperative analgesia — Patients will receive a patient-controlled intravenous or perineural catheter-based analgesia, depending on their preference and the anesthesiologist's indication.
  Other Names: PCA; PCIVA; PCCPNB; Patient-controlled continuous peripheral nerve block
Drug: Mepivacaine — Thirty milliliters of 1.5% (wt/vol) mepivacaine will be used for the sciatic nerve block.
  Other Names: Local Anesthetic; Carbocaine

SUMMARY:
This study was designed to assess whether the injection of local anesthetic into the nerve (intraneural), as opposed to around it (perineural), leads to longer anesthesia and analgesia of the leg.

Some reports of accidental intraneural injection mention an extremely long duration. When different drugs and doses were evaluated in a clinical trial of intraneural injection, a longer-than-expected duration was reported.

The investigators will compare the two types of injection using the same drug, so as to determine if there is an actual difference in duration.

DETAILED DESCRIPTION:
This randomized, controlled trial will investigate prospectively for differences in sensory and motor block duration after intra- or perineural injection of 1.5% (wt/vol) mepivacaine, a short-acting local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing non-emergent orthopedic procedure of knee, leg, foot with thigh tourniquet
* ASA Physical Status Class I-III
* Consenting to surgery under peripheral nerve block anesthesia (sciatic + femoral/saphenous block)

Exclusion Criteria:

* Unable to understand or communicate for the purpose of the study
* Exhibiting signs of neuropathy in the ipsilateral extremity
* Inability to satisfactorily image the sciatic nerve in the opinion of the attending anesthesiologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Differences in Time to Resolution of Sciatic Nerve Block | <12 h
  The time at which sensory and motor function of the sciatic nerve have recovered at least to the following criteria:
  * Sensory: patients feel discomfort when pricked with a thin needle (25G)
  * Motor: patients may move both toes and ankle, albeit with reduced strength
  This outcome measure will be examined by an investigator every 30-60 min and reported by patients as "time to return of sensation and movement". The investigator-reported value will be preferred if both are available.

SECONDARY OUTCOMES:
Block Onset Time | ≤30 min
  Time to onset of sciatic nerve anesthesia, defined as meeting at least the following criteria:
  * Sensory: does not feel pain or discomfort when pricked with a 25G needle.
  * Motor: able to slightly curl toes; unable to flex the ankle.
Success Rate of Anesthetic Nerve Blocks | ≤30 min
  The percentage of patients who attain the criteria for block success within 30 minutes of the injeciton.
  Investigators will also report the percentage of patients who successfully complete surgery without significant additional analgesia (see below); this will be defined as "clinical success rate."
Incidence and Prevalence of Neurologic Disturbances | 30 days
  Patients will be interviewed at ~4 h (block resolution visit), 7 days and (if necessary) at 30 days to assess for residual neurologic disturbances in the sciatic nerve territory.
  The incidence/prevalence of these phenomena will be noted.

OTHER OUTCOMES:
Extra- vs. Intraneural Minimum Electrical Stimulation Thresholds | (during the procedure)
  The minimum electrical nerve stimulation threshold will be recorded as a function of needle tip position.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Baciarello, MD, Principal Investigator — University of Parma
Locations (1):
- Anesthesia, Critical Care and Pain Medicine - University of Parma, Parma, PR, Italy

REFERENCES:
- [Background] Benhamou D, Blonski E, Levy P, Plessis E, Chalhoub V. Ultra-long duration of a peripheral nerve block: a possible consequence of intraneural (subepineural) local anaesthetic injection. Ann Fr Anesth Reanim. 2010 Jul-Aug;29(7-8):589-91. doi: 10.1016/j.annfar.2010.05.032. Epub 2010 Jul 13. PMID 20630694
- [Background] Nader A, Kendall MC, De Oliveira GS Jr, Puri L, Tureanu L, Brodskaia A, Asher Y, Parimi V, McCarthy RJ. A dose-ranging study of 0.5% bupivacaine or ropivacaine on the success and duration of the ultrasound-guided, nerve-stimulator-assisted sciatic nerve block: a double-blind, randomized clinical trial. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):492-502. doi: 10.1097/AAP.0b013e3182a4bddf. PMID 24108248